CLINICAL TRIAL: NCT06710548
Title: Randomized Trial of REVITALIZE: A Telehealth Intervention to Reduce Fatigue Interference Among Adults With Advanced Ovarian Cancer on PARP Inhibitors
Brief Title: REVITALIZE: RCT to Reduce Fatigue in Adults With Ovarian Cancer on PARP Inhibitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-105; R01CA289547 (NIH)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Advanced Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Cancer; PARP Inhibitor; Fatigue Related to Cancer Treatment; Fatigue in Cancer Survivors
Keywords: Ovarian Cancer; Advanced Ovarian Carcinoma; Advanced Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Fatigue related to cancer treatment; Fatigue in Cancer Survivors; PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1: REVITALIZE Intervention (Experimental): 120 participants will be randomized in a 1:1 fashion stratified by PARP inhibitor type and study site and will complete the following:
  1. Questionnaire upon enrollment.
  2. Use of a wireless pill bottle for PARP inhibitor medication.
  3. Eight weekly one-on-one intervention sessions with a coach via Zoom.
  4. Two booster sessions to reinforce intervention with a coach via Zoom.
  5. Questionnaires at 8, 13, 20, and 28 weeks.
  Interventions: Behavioral: REVITALIZE Intervention
- ARM 2: Educational Materials (Active Comparator): 120 participants will be randomized in a 1:1 fashion stratified by PARP inhibitor type and study site and will complete the following:
  1. Questionnaire upon enrollment.
  2. Use of wireless pill bottle for PARP inhibitor medication.
  3. Educational information on cancer survivorship, including management of fatigue.
  4. Questionnaires at 8, 13, 20, and 28 weeks.
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: REVITALIZE Intervention — A remotely delivered tele-health intervention to address cancer fatigue that is based on an acceptance-based approach. The intervention includes 8 one-on-one weekly sessions and 2 booster sessions with trained psychology doctoral students based at University of Colorado. Sessions will focus on fatigue education, Acceptance and Commitment Therapy (ACT) skills, and behavior changes. Wi-Fi enabled tablets and keyboards will be provided to participants if needed. All sessions will be conducted via the Zoom platform and will either be videotaped or audiotaped.
  Arms: ARM 1: REVITALIZE Intervention
Behavioral: Educational Materials — The educational materials arm will receive specialized cancer survivorship educational materials created by the National Cancer Institute
  Arms: ARM 2: Educational Materials

SUMMARY:
The purpose of this study is to see whether a supportive intervention (REVITALIZE) reduces fatigue and its impact on daily life and activities for participants with ovarian cancer taking PARP inhibitors.

The name of the study groups in this research study are:

1. REVITALIZE
2. Educational Materials

DETAILED DESCRIPTION:
This Phase 3 randomized controlled trial will evaluate the effect of a brief, acceptance-based tele-health intervention (REVITALIZE) vs. educational materials in participants with ovarian cancer who are taking poly-ADP ribose polymerase (PARP) inhibitors.

Participants will be randomized into one of two study groups: 1) REVITALIZE or 2) Educational Materials. Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, using a wireless pill bottle, and completing questionnaires.

Participation in this research study is expected to last about 7 months.

It is expected about 240 people will take part in this research study.

The National Cancer Institute is supporting this research by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) with ovarian, fallopian tube, or primary peritoneal cancers (hereafter ovarian cancer) who have completed primary therapy (surgery and chemotherapy).
* Treated with a PARP inhibitor as maintenance therapy for ≥2 months and plan to continue for at least 7 months.
* English-speaking.
* Mean fatigue severity level ≥4 on the first three items of the Fatigue Symptom Inventory.
* ECOG performance status of 0-2.
* Willing to use a wireless pill bottle for PARP inhibitor medication.

Exclusion Criteria:

* Untreated clinical condition or comorbid condition that pre-dates PARP inhibitor use and could explain fatigue, as evaluated by their treating oncologist.
* Patients with severe psychiatric conditions (e.g. untreated trauma unrelated to cancer, high or imminent suicidality) as evaluated by their treating oncologist, which require more intensive psychiatric treatment than the study can provide.
* Patients with cognitive conditions (e.g. dementia), determined by their treating oncologist, such that they could not provide informed consent or complete the study procedures.
* Inability to complete the first questionnaire within one week of consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Interference Score from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the 7-item Fatigue Interference subscale of the Fatigue Symptom Inventory (FSI). Items are rated on an 11-point scale (0 = no interference; 10 = extreme interference), with a total scores range of 0 to 70 with the higher score representing greater fatigue interference with daily life. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.

SECONDARY OUTCOMES:
Change in Fatigue Interference Score from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed by the 7-item Fatigue Interference subscale of the Fatigue Symptom Inventory (FSI). Items are rated on an 11-point scale (0 = no interference; 10 = extreme interference), with a total scores range of 0 to 70 with the higher score representing greater fatigue interference with daily life. The mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the Patient-Reported Outcome Measurement Information system (PROMIS) Cancer Fatigue Short Form 7a, a 7-item measure rated on a 5-point scale (1 "never" to 5 "always") with a total scores range of 7 to 35, and a higher score representing greater fatigue severity. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed by the Patient-Reported Outcome Measurement Information system (PROMIS) Cancer Fatigue Short Form 7a, a 7-item measure rated on a 5-point scale (1 "never" to 5 "always") with a total scores range of 7 to 35, and a higher score representing greater fatigue severity.The mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue Self-Efficacy Score from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the Fatigue Self-Efficacy Scale, a 7-item measure that is rated on a 4 point scale of 1 "No, I am convinced that this is not the case" to 4 "Yes, I am convinced of that." A total scores range would be 7 to 28 with a higher score representing greater belief in the ability to improve fatigue. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue Self-Efficacy Score from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed by the Fatigue Self-Efficacy Scale, a 7-item measure that is rated on a 4 point scale of 1 "No, I am convinced that this is not the case" to 4 "Yes, I am convinced of that." A total scores range would be 7 to 28 with a higher score representing greater belief in the ability to improve fatigueThe mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue Catastrophizing Score from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the Fatigue Catastrophizing Scale, a 10-item survey rated on a 5 point scale with answers ranging from 1 "Never True" to 5 "All of the time true." A total scores range would be 7 to 50 with a higher score representing greater participant catastrophizing about fatigue. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Fatigue Catastrophizing Score from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed by the Fatigue Catastrophizing Scale, a 10-item survey rated on a 5 point scale with answers ranging from 1 "Never True" to 5 "All of the time true." A total scores range would be 7 to 50 with a higher score representing greater participant catastrophizing about fatigue. The mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Participant Sleep Disturbance from Baseline to 8 weeks (Arms 1 and 2) | 8 weeks
  Assessed by the PROMIS Sleep Disturbance Short Form 8a, an 8-item survey rated on a 5 point scale with answers ranging from (1 'Very Good' to 5 'Very Poor' or 1 'Very Much' to 5 'Not At All'), where lower scores represent less disturbance.
Change in Participant Sleep Disturbance from Baseline to 13 weeks (Arms 1 and 2) | 13 weeks
  Assessed by the PROMIS Sleep Disturbance Short Form 8a, an 8-item survey rated on a 5 point scale with answers ranging from (1 'Very Good' to 5 'Very Poor' or 1 'Very Much' to 5 'Not At All'), where lower scores represent less disturbance.
Change in Participant Sleep Disturbance from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the PROMIS Sleep Disturbance Short Form 8a, an 8-item survey rated on a 5 point scale with answers ranging from (1 'Very Good' to 5 'Very Poor' or 1 'Very Much' to 5 'Not At All'), where lower scores represent less disturbance.
Change in Quality of Life Score from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed by the PROMIS Global Health 10, a 10-item measure of physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, and ability to carry out usual social activities and roles, pain, fatigue and overall quality of life. Answers are rated on a 5-point scale (1 "Poor" to 5 "Excellent"; 1 "Not at all" to "Completely", where higher scores represents better participant well-being. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Quality of Life Score from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed by the PROMIS Global Health 10, a 10-item measure of physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, and ability to carry out usual social activities and roles, pain, fatigue and overall quality of life. Answers are rated on a 5-point scale (1 "Poor" to 5 "Excellent"; 1 "Not at all" to "Completely", where higher scores represents better participant well-being. The mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Emotional Distress: Anxiety Symptoms from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed using the Generalized Anxiety Disorder 7-Item (GAD-7), which is a reliable and validated self-report measure to assess anxiety symptoms. For the GAD-7, respondents rated how often they have been bothered by 7 anxiety symptoms over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. Respondents also answer a question to assess the duration of their anxiety symptoms. The scale is scored 0-21, where 0-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and scores >15 is severe anxiety. Using a cut-off of 8 the GAD-7 has a sensitivity of 92% and specificity of 76% for diagnosis generalized anxiety disorder.
Emotional Distress: Anxiety Symptoms from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed using the Generalized Anxiety Disorder 7-Item (GAD-7), which is a reliable and validated self-report measure to assess anxiety symptoms. For the GAD-7, respondents rated how often they have been bothered by 7 anxiety symptoms over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. Respondents also answer a question to assess the duration of their anxiety symptoms. The scale is scored 0-21, where 0-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and scores >15 is severe anxiety. Using a cut-off of 8 the GAD-7 has a sensitivity of 92% and specificity of 76% for diagnosis generalized anxiety disorder.
Emotional Distress: Depressive Symptoms from Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Assessed using 8-item Patient Health Questionnaire (PHQ-8), which is a reliable and validated self-report measure to assess depressive symptoms. For the PHQ-8, respondents rated how often they have been bothered by 8 symptoms of depression over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. The scale is totaled (range 0-24) where total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Emotional Distress: Depressive Symptoms from Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Assessed using 8-item Patient Health Questionnaire (PHQ-8), which is a reliable and validated self-report measure to assess depressive symptoms. For the PHQ-8, respondents rated how often they have been bothered by 8 symptoms of depression over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. The scale is totaled (range 0-24) where total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Poly-ADP Ribose Polymerase (PARP) Inhibitor Adherence Rate From Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Calculated as the percentage of daily doses taken per 30-day month (% days Wisepill is opened once for each dose prescribed that day/ 30), using recommended methods for Wisepill pillbox data preparation and analysis. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
PARP Inhibitor Adherence Rate From Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Calculated as the percentage of daily doses taken per 30-day month (% days Wisepill is opened once for each dose prescribed that day/ 30), using recommended methods for Wisepill data preparation and analysis. The mean change from baseline to the follow up time point (28 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
PARP Inhibitor Non-Persistence From baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  Defined as Wisepill pillbox monitoring detecting that a participant stops taking medication entirely from Baseline through 20 weeks follow up. The measure will be quantified as yes/no binary outcomes with yes = any dose delay [or interruption] from baseline to 20 week follow up and no = no dose delay [or interruption] from baseline to 20 week follow up. The proportion and a corresponding 0.95 asymptotic confidence interval will be computed.
PARP Inhibitor Non-Persistence From baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  Defined as Wisepill pillbox monitoring detecting that a participant stops taking medication entirely from Baseline through 28 week follow up. The measure will be quantified as yes/no binary outcomes with yes = any dose delay [or interruption] from baseline to 28 week follow up and no = no dose delay [or interruption] from baseline to 28 week follow up. The proportion and a corresponding 0.95 asymptotic confidence interval will be computed.
PARP Inhibitor Regimen by Medical Chart Abstraction From Baseline to 20 weeks (Arms 1 and 2) | 20 weeks
  PARP inhibitor treatment will be measured via medical chart abstraction. The measure will be quantified as yes/no binary outcomes with yes = any dose delay [or interruption] from baseline to 4 month follow up and no = no dose delay [or interruption] from baseline to 20 week follow up. The proportion and a corresponding 0.95 asymptotic confidence interval will be computed.
PARP Inhibitor Regimen by Medical Chart Abstraction From Baseline to 28 weeks (Arms 1 and 2) | 28 weeks
  PARP inhibitor treatment will be measured via medical chart abstraction. The measure will be quantified as yes/no binary outcomes with yes = any dose delay [or interruption] from baseline to 28 week follow up and no = no dose delay [or interruption] from baseline to 28 week follow up. The proportion and a corresponding 0.95 asymptotic confidence interval will be computed.
Change in Value-Aligned Behavior Score From Baseline to 8 weeks (Arms 1 and 2) | 8 weeks
  Mechanism measure assessed by the Valuing Questionnaire (VQ), a 10-item survey that measures value aligned behaviors in the past week. Responses are measured on a 6 point scale with answers ranging from 0 "not at all true" to 6 "completely true" with a total scores range of 0 to 60, and a higher score representing greater value to behavior alignment. The mean change from baseline to the follow up time point (8 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Value-Aligned Behavior Score From Baseline to 13 weeks (Arms 1 and 2) | 13 weeks
  Mechanism measure assessed by the Valuing Questionnaire (VQ), a 10-item survey that measures value aligned behaviors in the past week. Responses are measured on a 6 point scale with answers ranging from 0 "not at all true" to 6 "completely true" with a total scores range of 0 to 60, and a higher score representing greater value to behavior alignment. The mean change from baseline to the follow up time point (13 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval.
Change in Acceptance and Cognitive Defusion from Baseline to 8 weeks (Arms 1 and 2) | 8 weeks
  Mechanism measure assessed by the Experiences Questionnaire Decentering Scale, a 13-item survey that measures acceptance and cognitive defusion. Responses are measured on a 5-point Likert scale from 1 'Never' to 5 'All the time,' range from 13 to 65, and a higher representing greater acceptance and defusion.
Change in Acceptance and Cognitive Defusion from Baseline to 13 weeks (Arms 1 and 2) | 13 weeks
  Mechanism measure assessed by the Experiences Questionnaire Decentering Scale, a 13-item survey that measures acceptance and cognitive defusion. Responses are measured on a 5-point Likert scale from 1 'Never' to 5 'All the time,' range from 13 to 65, and a higher representing greater acceptance and defusion.
Acceptability of Intervention (Arms 1 and 2) | 13 weeks
  Assessed by the Acceptability of Intervention Measure, a 4-item survey rated on a 5 point scale with answers ranging from 1 'Completely disagree' to 5 'Completely agree.' Total scores range from 4 to 20, with the higher number indicating greater satisfaction. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval
Acceptability of Intervention (Arms 1 and 2) | 20 weeks
  Assessed by the Acceptability of Intervention Measure, a 4-item survey rated on a 5 point scale with answers ranging from 1 'Completely disagree' to 5 'Completely agree.' Total scores range from 4 to 20, with the higher number indicating greater satisfaction. The mean change from baseline to the follow up time point (20 weeks) will be computed using a two-sample t-test with a 0.95 confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A Wright, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute; Joanna J Arch, PhD, Principal Investigator — University of Colorado, Boulder
Locations (6):
- United States (6):
  - University of Colorado Cancer Center-Anschutz, Aurora, Colorado
  - University of Colorado Boulder, Boulder, Colorado
  - Massachusetts General Hospital-Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Cancer Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu